CLINICAL TRIAL: NCT03592264
Title: A Phase I/II Study of OBI-3424 in Subjects with Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Little evidence of clinical activity in tumor types enrolled
Sponsor: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OBI-3424-001
Record Dates: First submitted 2018-05-21; First posted 2018-07-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor; Pancreatic Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation phase (Experimental): OBI-3424 (1.0 mg/m^2 to 14.0 mg/m^2) will be administered by IV infusion on Days 1 and 8 of each 21-day cycle or Day 1 of each 21-day cycle to determine the MTD and RP2D with a classic 3+3 dose escalation design.
  Interventions: Drug: OBI-3424
- Cohort expansion phase (Experimental): OBI-3424 (12 mg/m^2) will be administered by IV infusion on Day 1 of each 21-day cycle.
  Interventions: Drug: OBI-3424

INTERVENTIONS:
Drug: OBI-3424 — liquid formulation for Intravenous infusion

SUMMARY:
A first-in-human open-label, Phase I/II study to evaluate the safety, tolerability, MTD/RP2D, PK, and preliminary efficacy of OBI-3424 administered as a single agent.

ELIGIBILITY:
Inclusion Criteria (all subjects):

1. At least 18 years of age
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC)
3. Recovered from toxicities of prior therapy to Grade 0 or 1
4. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) criteria
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Acceptable liver function:

   1. Bilirubin ≤1.5 × institutional ULN
   2. AST and ALT ≤3.0 × ULN, or ≤5.0 × ULN for subjects with liver involvement
7. Acceptable renal function:

   a. Creatinine clearance >30 mL/min according to the Cockcroft-Gault formula
8. Acceptable hematologic status (without hematologic support, other than red blood cell transfusion):

   1. ANC ≥1500 cells/μL
   2. Platelet count ≥100,000/μL
   3. Hemoglobin ≥9.0 g/dL (prior packed red blood cell transfusion or erythropoietin support is allowed).
9. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation.

   Dose Escalation Phase Subjects Only (Inclusion Criteria):
10. Histologically or cytologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
11. Tumor progression after most recent therapy

    Expansion Phase Subjects Only (Inclusion Criteria):
12. Available tumor tissue, either archival or fresh (fresh preferred).
13. For treatment, an AKR1C3 IHC H-score of ≥ 100 using a validated IHC assay in one of the following tumor types to be enrolled in the respective cohort:

    1. Cohort A: Pancreatic Adenocarcinoma
    2. Cohort B: Basket (any solid tumor type other than pancreatic adenocarcinoma)

Exclusion Criteria:

1. Prior radiotherapy to more than 25% of the bone marrow
2. Symptomatic brain metastases, unless previously treated and well controlled for at least 4 weeks after central nervous system (CNS)-directed treatment as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]) during the Screening Period. Patients with known leptomeningeal disease are excluded.
3. Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancers whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the current study
4. Patients with hepatocellular carcinoma (applies to Expansion Phase only)
5. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
6. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
7. Treatment with radiation therapy, surgery, chemotherapy, targeted therapies or hormones within 3 weeks prior to study entry (6 weeks for nitrosoureas or mitomycin C)
8. Concomitant use of strong CYP3A4 inhibitors/inducers
9. Concomitant use of naproxen within a 48-hour window before and after OBI-3424 dosing
10. Females who are pregnant or breast-feeding
11. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
12. Unwillingness or inability to comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Adverse events will be noted as it occurs. Timeframe for measure begins after first administration of study drug until 30 days after last dose of study drug. Study duration defined as up to 2 years from the first dose.
  Adverse events will be graded according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Assess safety changes in electrocardiogram (ECG) | Day 1 Cycles 1 and 2 (each cycle is 21 days)
  Resting 12-lead ECGs will be obtained from all subjects' pre-OBI-3424 infusion and within 15 minutes post-OBI-3424 infusion in order to assess any impact OBI-3424 may have on the QT interval as assessed by the Fridericia's Correction Formula (QTcF).
Assess safety changes of body weight. | Day 1 of each cycle (there are 34 cycles; 21 days for each cycle)
  If during treatment a subject's body weight changes by >10%, the dose should be adjusted.
Number of participants with dose limiting toxicities (DLTs) | Throughout Cycle 1 (21 days for each cycle)
  A DLT is defined as the occurrence of Grade 3/4 adverse events within the first cycle (the first 21 days) of treatment that are considered by the investigator to be at least possibly related to OBI-3424.
Define the Recommended Phase 2 Dose (RP2D) | Days 1 and 8 of each cycle (all 34 cycles and there are 21 days for each cycle)
  Determination of the MTD, based on the frequently of DLTs observed in Cycle 1 in subjects recruited to the Dose Escalation Phase.
Pharmacokinetics (PK) - Time to maximum concentration (Tmax) | Days 1 and 8 of Cycle 1 (first cycle of 34 cycles and there are 21 days for each cycle)
  Tmax of OBI-3424 and OBI-2660 will be computed for each subject where possible.
PK - Maximum peak plasma concentration (Cmax) | Days 1 and 8 of Cycle 1 (first cycle of 34 cycles and there are 21 days for each cycle)
  Cmax of OBI-3424 and OBI-2660 will be computed for each subject where possible.
PK - The magnitude of the slope of the linear regression of the log concentration vs. time profile during the terminal phase (Kel) | Days 1 and 8 of Cycle 1 (first cycle of 34 cycles and there are 21 days for each cycle)
  Kel of OBI-3424 and OBI-2660 will be computed for each subject where possible.
PK - Half-life (T1/2) | Days 1 and 8 of Cycle 1 (first cycle of 34 cycles and there are 21 days for each cycle)
  T1/2 computed as ln (2)/Kel of OBI-3424 and OBI-2660 will be computed for each subject where possible.
PK - Area under the concentration-time curve (AUClast) | Days 1 and 8 of Cycle 1 (Cycle 1 is 21 days)
  AUClast from Hour 0 through the last quantifiable concentration time (LQCT), where LQCT is the time at which the last sample with a quantifiable concentration was drawn

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia Tsimberidou, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Scripps Clinic Torrey Pines, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tsimberidou AM, Verschraegen CF, Wesolowski R, Shia CS, Hsu P, Pearce TE. Phase 1 dose-escalation study evaluating the safety, pharmacokinetics, and clinical activity of OBI-3424 in patients with advanced or metastatic solid tumors. Br J Cancer. 2023 Aug;129(2):266-274. doi: 10.1038/s41416-023-02280-4. Epub 2023 May 12. PMID 37173365